CLINICAL TRIAL: NCT01750723
Title: Basic Research on Acetazolamide´s Headache Inducing Characteristics and Effects on the Cerebral Arteries and Blood Flow in a Humane Experimental Headache Model
Brief Title: Acetazolamide's Headache Inducing Characteristics and Effects on the Cerebral Arteries and Blood Flow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Nanna Arngrim, MD, medical doctor, Danish Headache Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H-3-2012-137
Record Dates: First submitted 2012-12-11; First posted 2012-12-17 (Estimated); Last update posted 2013-07-09 (Estimated); Status verified 2013-07

CONDITIONS: Headache; Migraine
Keywords: Acetazolamide; Headache; Migraine
MeSH Terms: conditions — Headache; Migraine Disorders | interventions — Acetazolamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acetazolamide (Active Comparator): Acetazolamide 1 g in 10 ml saline, i.v. infusion
  Interventions: Drug: Acetazolamide
- Saline (Placebo Comparator): Saline, 10 ml i.v. infusion

INTERVENTIONS:
Drug: Acetazolamide — 1 g diluted in 10 ml saline, i.v. bolus injection.
  Other Names: Diamox
  Arms: Acetazolamide

SUMMARY:
In this study the investigators will research the hypothesis that the drug Acetazolamide induce headache and dilation of cerebral arteries and increase the cerebral blood flow in the areas of the brain supplied by these arteries.

DETAILED DESCRIPTION:
To investigate headache score and accompanying symptoms during and after infusion of acetazolamide.

With magnetic resonance imaging the investigators will investigate changes in regional cerebral blood flow (rCBF) in the area supplied by middle cerebral artery (MCA), diameter of MCA, the Internal carotic artery (ICA), the superficial temporal artery (STA) and the Medial Meningeal artery (MMA).

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Aged 18-40
* 50-100 kg
* Fertile women must use safe contraceptives (IUD, oral contraceptives, surgical sterilisation and long lasting gestagen.

Exclusion Criteria:

* Tension type headache more than once/month
* Other primary headaches
* Daily medication except contraceptives
* Drug taken within 4 times the halflife for the specific drug except contraceptives
* Pregnant or lactating women
* Exposure to radiation within the last year
* Headache within the last 24 hours before start of trial
* Hypertension
* Hypotension
* Respiratory or cardiac disease

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-12; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Headache scores | 24 h
  Comparison between Acetazolamide and placebo (saline).

SECONDARY OUTCOMES:
Artery circumference | Baseline, 30 min and 60 min
  Acetazolamide induced changes in intracranial artery circumference before and after infusions.
Cerebral blood flow | Baseline, 30 and 60 min.
  Acetazolamide induced changes in cerebral blood flow.

CONTACTS AND LOCATIONS:
Overall Officials: Nanna Arngrim, MD, Principal Investigator — Danish Headache Center
Locations (2):
- Denmark (2):
  - Danish Headache Center, Copenhagen, Glostrup
  - Department of Neurology, Copenhagen, Glostrup